CLINICAL TRIAL: NCT03758885
Title: A Phase 3, Double-blind, Randomized, Placebo-controlled Study to Assess the Safety and Efficacy of a Single Oral Administration of Nolasiban to Increase On-going Pregnancy Rate Following Fresh Single Blastocyst Transfer Resulting From IVF
Brief Title: Study of Nolasiban to Increase Pregnancy Rates in Women Undergoing IVF
Acronym: IMPLANT4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ObsEva SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-OBE001-010
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2020-09

CONDITIONS: Infertility
Keywords: IVF; ICSI; ART; ET
MeSH Terms: conditions — Infertility | interventions — nolasiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nolasiban 900 mg (Experimental): Nolasiban dispersible tablets for single oral administration
  Interventions: Drug: Nolasiban
- Placebo (Placebo Comparator): Placebo dispersible tablets for single oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nolasiban — Nolasiban single oral administration
  Arms: Nolasiban 900 mg
Drug: Placebo — Placebo single oral administration
  Arms: Placebo

SUMMARY:
The primary objective of this study is to confirm the efficacy of a single oral 900 mg dose of nolasiban versus placebo to increase the ongoing clinical pregnancy rate at 10 weeks post-embryo transfer (ET) day.

DETAILED DESCRIPTION:
The study is a prospective, randomised, parallel group, double-blind, placebo-controlled, Phase 3 study to confirm the efficacy and the safety of nolasiban versus placebo to increase pregnancy and live birth rates in 820 women undergoing fresh single blastocyst transfer following in vitro fertilisation (IVF) or intra-cytoplasmic sperm injection (ICSI).

ELIGIBILITY:
Inclusion Criteria:

* Indicated for IVF/ICSI in the context of assisted reproductive technology (ART)
* Follow a gonadotropin releasing hormone (GnRH) antagonist protocol, single injection of human chorionic gonadotropin (hCG) for triggering final follicular maturation and luteal support with vaginal micronized progesterone.
* Single fresh D5 embryo transfer

Exclusion Criteria:

* Frozen-thawed embryo transfer
* Donor egg in the current transfer
* More than 20 oocytes in the current controlled ovarian hyperstimulation (COH) cycle
* Serum P4 greater than 1.5 ng/mL prior to hCG administration

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 820 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy with fetal heart beat at 10 weeks | 10 weeks post ET day
  Ongoing pregnancy defined as an intra-uterine pregnancy with fetal heart beat at 10 weeks post embryo transfer day

SECONDARY OUTCOMES:
Live birth | 24 to 40 weeks of gestation
  Live birth after 24 weeks of gestation
Clinical pregnancy at 6 weeks post ET day | 6 weeks post ET
  Clinical pregnancy defined as intra-uterine pregnancy with fetal heart beat at 6 weeks post-ET day
Pregnancy rate at 14 days post Oocyte Pick-up (OPU) | 14 days post OPU
  Positive blood pregnancy test at 14 days post OPU day
Pregnancy loss | 6 weeks post ET to 24 weeks gestation
  Pregnancy loss at 6 or 10 weeks after ET and before 24 weeks of gestation
Plasma concentrations of nolasiban | 3.5 hours, 5 hours and at 7 hours (latest 72 hours) after nolasiban administration
  Plasma concentrations of nolasiban after administration

OTHER OUTCOMES:
Adverse events | Through study completion, up to 11 months
  Treatment emergent adverse events frequency and severity
Neonatal assessments | Birth of infant until 28 days
  Incidence of any malformation or any significant morbidity during the neonatal period
Ages and Stages Questionnaires® (ASQ-3™) 6 and 12 month Questionnaire | 6 and 12 months after term
  Screening questionnaire composed of 30 questions completed by the parent. Questions are divided into five areas: communication, gross motor, fine motor, problem solving and personal-social. Parents respond yes, sometimes and not yet to questions, these are converted to points 10, 5 and 0 for scoring and are totalled for each developmental area. These 5 area scores are compared with empirically derived cutoff points.

CONTACTS AND LOCATIONS:
Locations (50):
- Belgium (4):
  - Site 1001, Brussels
  - Site 1002, Brussels
  - Site 1003, Brussels
  - Site 1004, Brussels
- Canada (4):
  - Site 1404, Burnaby
  - Site 1401, Montreal
  - Site 1402, Toronto
  - Site 1403, Toronto
- Czechia (10):
  - Site 1107, Olomouc
  - Site 1101, Prague
  - Site 1102, Prague
  - Site 1103, Prague
  - Site 1104, Prague
  - Site 1105, Prague
  - Site 1108, Prague
  - Site 1110, Prague
  - Site 1109, Teplice
  - Site 1106, Zlín
- Denmark (4):
  - Site 1204, Copenhagen
  - Site 1205, Herlev
  - Site 1202, Hvidovre
  - Site 1203, Skive
- Estonia (3):
  - Site 1302, Tallinn
  - Site 1301, Tartu
  - Site 1303, Tartu
- Germany (6):
  - Site 1504, Berlin
  - Site 1506, Berlin
  - Site 1505, Bielefeld
  - Site 1501, Heidelberg
  - Site 1502, Lübeck
  - Site 1503, Marburg
- Hungary (3):
  - Site 1601, Budapest
  - Site 1603, Budapest
  - Site 1602, Tapolca
- Poland (6):
  - Site 1703, Bialystok
  - Site 1705, Bialystok
  - Site 1702, Katowice
  - Site 1701, Krakow
  - Site 1704, Szczecin
  - Site 1706, Warsaw
- Russia (4):
  - Site 1901, Moscow
  - Site 1905, Moscow
  - Site 1904, Samara
  - Site 1902, Yekaterinburg
- Spain (6):
  - Site 1805, Barcelona
  - Site 1808, Barcelona
  - Site 1809, Leioa
  - Site 1804, Madrid
  - Site 1807, Madrid
  - Site 1811, Seville

REFERENCES:
- [Derived] Griesinger G, Blockeel C, Pierzynski P, Tournaye H, Visnova H, Humberstone A, Terrill P, Pohl O, Garner E, Donnez J, Loumaye E. Effect of the oxytocin receptor antagonist nolasiban on pregnancy rates in women undergoing embryo transfer following IVF: analysis of three randomised clinical trials. Hum Reprod. 2021 Mar 18;36(4):1007-1020. doi: 10.1093/humrep/deaa369. PMID 33534895